CLINICAL TRIAL: NCT03981276
Title: Phenotypes, Biomarkers and Pathophysiology in Hereditary Spastic Paraplegias and Related Disorders
Acronym: HSP-PBP
Status: Recruiting | Type: Observational
Sponsor: Dr. Rebecca Schule (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government); German Center for Neurodegenerative Diseases (DZNE) (Other)
Responsible Party: Sponsor-Investigator, Dr. Rebecca Schule, Principal Investigator, Leading Consultant, University Hospital Tuebingen
Organization: University Hospital Tuebingen (Other)
Other Study IDs: HSP-PBP; 01GM1905 (Other Grant/Funding Number: Bundesministerium für Bildung und Forschung (BMBF))
Record Dates: First submitted 2019-06-04; First posted 2019-06-10 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Hereditary Spastic Paraplegia
Keywords: Hereditary Spastic Paraplegia; Biomarker; Genetic etiology; Molecular mechanisms
MeSH Terms: conditions — Spastic Paraplegia, Hereditary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Biospecimen Retention: Samples With DNA — optional biosample collection including blood (DNA, serum, plasma, RNA, PBMC), urine, CSF, skin biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Primary participant:: Participants affected by hereditary spastic paraplegia (HSP) or a phenotypically related disorder Primary participants will be followed at annual intervals. The workup includes clinical, imaging, sensor-based, patient/observer reported and molecular outcome parameters and biosampling.
  Participants with unknown genetic diagnosis may receive genetic testing including whole exome or whole genome sequencing and other OMICS techniques.
  Interventions: Other: Clinical rating scale to measure disease severity and progression; Diagnostic Test: Next-Gen Sequencing (NGS)
- Secondary participant/ First or second-degree: First or second degree unaffected family members of primary participants. Secondary participants may undergo the same study procedures as primary participants.
  Interventions: Diagnostic Test: Next-Gen Sequencing (NGS)
- Unrelated healthy control: Unrelated healthy controls Healthy controls may undergo the same study procedures as primary participants.
  Interventions: Diagnostic Test: Next-Gen Sequencing (NGS)

INTERVENTIONS:
Other: Clinical rating scale to measure disease severity and progression — A 13-item scale to rate functional impairment occurring in pure forms of spastic paraplegia (SP). Additional symptoms constituting a complicated form of SP are recorded in an inventory.
  Other Names: Spastic Paraplegia Rating Scale (SPRS)
  Groups: Primary participant:
Diagnostic Test: Next-Gen Sequencing (NGS) — Whole Genome Sequencing, Whole Exome Sequencing, Transcriptomics, Proteomics, Metabolomics

SUMMARY:
The aim of this study is to determine the clinical spectrum and natural progression of Hereditary Spastic Paraplegias (HSP) and related disorders in a prospective multicenter natural history study, identify digital, imaging and molecular biomarkers that can assist in diagnosis and therapy development and study the genetic etiology and molecular mechanisms of these diseases.

DETAILED DESCRIPTION:
The investigators will perform a registry-based standardized prospective Natural History Study (NHS) in HSPs and related disorders. Participants will be seen annually. At study visits a standardized clinical examination will be performed including application of clinical rating scales (selection of rating scales may vary depending on the individual phenotype and specific genotype); data will be entered into a clinical database (HSP Registry; https://www.hsp-registry.net). At all study visits, patients will be asked to donate biosamples; biomaterial collection is optional and participants can elect to participate in sampling of blood, urine, CSF, and/or a skin biopsy.

Optionally, additional examinations may be performed including imaging, quantitative movement analysis, neuropsychological examinations, analysis of patient or observer reported outcomes and OMICS analysis to characterize molecular biomarkers.

In participants without a genetic diagnosis, next generation sequencing may be performed.

ELIGIBILITY:
Inclusion criteria:

* One of the following:

  1. Primary participant: Clinical or genetic diagnosis of HSP or a related disorder
  2. Secondary participant: Unaffected family member (1st or 2nd degree relative) of primary participant (with the above-mentioned restrictions for special populations) able to give informed consent
  3. Unrelated healthy control able to give informed consent

     AND
* Written informed consent

AND

- Participants are willing and able to comply with study procedures

Exclusion criteria:

* Missing informed consent of primary or secondary participant/ healthy control/ legal representatives
* For controls: evidence of a neurodegenerative disease or movement disorders; inability to give informed consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Probands with a clinical or genetic diagnosis of an HSP and related disorders including pre-manifest individuals will be primarily enrolled in this study (primary participants).
  Additionally, unaffected family members of primary participants will be enrolled if they are of legal age (>= 18 years) and able to give informed consent (secondary participants).
  Unaffected minors will only be enrolled under special circumstances as detailed in paragraph 5.1 (Special Populations - Unaffected minors).
  Lastly, healthy unrelated controls will be enrolled; these are necessary to contrast unspecific, gender- or age-related findings to disease specific findings.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2019-10-14 (Actual); Primary Completion 2039-08 (Estimated); Study Completion 2041-08 (Estimated)

PRIMARY OUTCOMES:
Change from baseline of Spastic Paraplegia Rating Scale (SPRS) total score at 2 years | up to 2 years
  Disease severity will be assessed by application of the Spastic Paraplegia Rating Scale (SPRS), a clinical rating scale measuring disease severity in Hereditary Spastic Paraplegia (Schüle et al. Neurology 2006). The SPRS contains 13 items, each ranging from 0 to 4 points. The total score is calculated as the sum of all items, yielding a range for the total score between 0 and 52. Hereby, higher SPRS total scores indicate more severe disease.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Schüle, PD Dr., Principal Investigator — University Hospital Tübingen
Locations (13):
- University Innsbruck, Innsbruck, Austria
- Germany (11):
  - German Center for Neurodegenerative Diseases (DZNE) Bonn, Bonn
  - University of Erlangen, Erlangen
  - University Medicine Essen, Essen
  - University Göttingen, Göttingen
  - University Heidelberg, Heidelberg
  - University of Lübeck, Lübeck
  - German Center for Neurogedenerative Diseases (DZNE) Magdeburg, Magdeburg
  - German Center for Neurodegenerative Diseases (DZNE) München, München
  - University of Regensburg, Regensburg
  - German Center for Neurodegenerative Diseases (DZNE) Rostock, Rostock
  - University of Tübingen and German Center for Neurodegenerative Diseases (DZNE) Tübingen, Tübingen
- IRCCS Medea Scientific Institute, Conegliano-PIeve di Soligo Research Centre, Pieve di Soligo, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Website of the TreatHSP consortium — http://treathsp.net
- See also: Website of the HSP Registry — http://hsp-registry.net